CLINICAL TRIAL: NCT06025019
Title: Effectiveness of Parent-based Electronic Health (eHealth) Intervention on Preschoolers' Physical Activity, Dietary Behaviors, and Sleep Problems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Beijing Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HKBU21481504ZP
Record Dates: First submitted 2023-07-09; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-05

CONDITIONS: Healthy Lifestyle; Physical Activity; Dietary Behaviors; Sleep
Keywords: physical activity; dietary behaviors; sleep; parent-based intervention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This study is a two parallel-group, single-blinded randomized controlled trial designed to promote preschoolers' PA, and DB, and reduce sleep problems by providing parents with relevant health information through the eHealth modality. The two arms comprise (1) eHealth intervention and (2) control group.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic Health (eHealth) (Experimental): Participants allocated to the eHealth intervention group will be delivered the evidence-based information and interactive components via social media (i.e., WeChat, similar to WhatsApp; and TikTok/Douyin, similar to YouTube). The interactive components include game, push notification, social rapport, influence agent, goal setting and personalized feedback.
  Interventions: Behavioral: parent-based Electronic Health intervention
- Control group (No Intervention): Participants allocated to the control group will be delivered printed evidence-based educational materials on standard recommendations for PA, diet, and sleep, without interactive components.

INTERVENTIONS:
Behavioral: parent-based Electronic Health intervention — The eHealth intervention comprises 12 modules on three interaction modules related to physical activity, dietary behavior, and sleep. The intervention groups will be invited to a "WeChat group". A 3-minute video (made on the TikTok APP) will be sent to each WeChat group. Based upon the social media studies recommendation, five to nine members in a group will produce the desirable group interactive effect. Therefore, the present study allocates eight parents to one WeChat group. In total, there will be 26 groups (206 parents) according to the sample size calculation. Consistent with Social Cognitive THeory, the content of each module will follow the four steps: 1. Attention (Read educational material and watch TikTok/Douyin video (less than 3 minutes). 2.Retention (parental interaction). 3.Reproduction (Set goals and conduct behaviors). 4.Motivation (feedback and making changes).
  Arms: Electronic Health (eHealth)

SUMMARY:
Background: Preschoolers' lifestyles have become physically inactive and sedentary, their eating habits unhealthy, and their sleep routines increasingly disturbed. Parental involvement appears to be crucial to combat unhealthy lifestyle of preschoolers. Because of recognized barriers of traditional face-to-face interventions (such as time commitment for parents), easy access and lower costs make electronic health (eHealth) interventions appealing. Previous studies that examined the effectiveness of parent-based eHealth on preschooler's (physical activity) PA, dietary behaviors (DB), and sleep have either emphasized on one variable or failed to balance the dosage of PA, diet, and sleep modules or consider the intervention sequence during the intervention period and there is an acknowledged gap in parent-based eHealth interventions which target preschoolers raised in Chinese cultural contexts.

Objective: This study aims to investigate the effectiveness of parent-based eHealth intervention on Chinese preschoolers' PA, DB, and sleep problems.

Methods: This two-arm parallel randomized controlled trial comprises a 12-week intervention with a 12-week follow-up. 206 parent-child dyads will be randomized to either eHealth intervention group or control group. Participants allocated to the eHealth intervention will receive 12 interactive modules on PA, DB, and sleep, with each module rot on a weekly basis to reduce the sequence effect on variable outcomes. The intervention is grounded upon Social Cognitive Theory and will be delivered through social media, where parents can obtain valid and updated educational information, social rapport, and interact with other group members and facilitators. Participants in the control group will receive weekly brochures on PA, DB, and sleep recommendations from the kindergarten teachers, but they will not receive any interactive components. Data will be collected at baseline, 3 months, and 6 months. The primary outcome will be the preschooler's physical activity. The secondary outcomes will be the preschooler's dietary behaviors, preschooler's sleep duration, and preschooler's sleep problems, parent's PA, parenting style, and parental feeding style.

Significance of this study: The parent-based eHealth intervention has potential to overcome the aforementioned barriers of face-to-face interventions, which will offer a novel approach for promoting healthy lifestyle of preschoolers. If found to be efficacious, the prevalence of unhealthy lifestyles among preschoolers may be alleviated at a low cost, which not only has a positive influence on the health of the individual and the well-being of the family but also reduces the financial pressure on society to treat diseases caused by poor lifestyle habits.

ELIGIBILITY:
Inclusion Criteria:

1. Parents are beyond 21 years old and have 4-6-year-old children. Selection of this child's age range was based on two factors. First of all, the age ranges from 4 to 6 have been found to be a strong predictor of future health. Secondly, a significant barrier to healthy DB is food neophobia, commonly known as picky or fussy eating, a reluctance, fear, or refusal to have new foods that is common in young children aged from 4 to 7.5 years.
2. Parental commitment to participate in the overall 6-month intervention.
3. Parents have access to mobile technology.
4. Parents and children must be healthy (refer to a state of physical, mental, social, intellectual, and emotional well-being and the absence of disease) and can participate in normal PA.
5. Parents must reside with participating child for at least four days a week (for the children to be adequately exposed to the intervention that parents may implement).

Exclusion Criteria:

1. if they meet the WHO criteria for preschool age children in terms of PA (i.e., 180 minutes of in a variety of PA at any intensity, of which 60 minutes is MVPA), sedentary behaviors (i.e., no more than 1 hour at a time being sedentary such as sit in car, no more than 1 hour per day in screen time such as TV, phone, and computer), DB (such as daily salt intake should be less than 5g), and sleep time (i.e., over 10 hours good quality sleep including nap, with regular sleep and wake time).
2. they diagnosed with neurological or physically disable and children who have a parent suffering from a serious physical or psychological disease making the study too demanding for the family will be excluded from the study.
3. if they have special dietary requirements or allergies that would necessitate the tailoring intervention or that may be adversely affected by the intervention. Eligible participants will be required to provide informed consent by completing a written consent form after reading the participant information.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 512 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Change of preschoolers' physical activity | Through study completion, 24 weeks
  Preschoolers' PA will be assessed baseline, at the end of 12-week post-intervention, and at the end of 12-week follow-up, using Garmin vivofit Jr 3 Fitness Tracker for Kids, which is a wrist-wear watch designed specifically for children from 4 to 9 years old to track PA in terms of steps and moderate-to-vigorous physical activity (MVPA) in minutes per day but not energy expenditure. This device has shown to be valid and accurate in assessing PA in preschoolers.

SECONDARY OUTCOMES:
Change of preschoolers' dietary behaviors | Through study completion, 24 weeks
  Preschoolers' dietary behaviors will be assessed at baseline, at the end of 12-week post-intervention, and at the end of 12-week follow-up, using Children's Eating Behavior Questionnaire (CEBQ), which has been examined the validity in Chinese preschool-age children. The scales have high internal consistency reliability (range .72-.91) and test-retest reliability (range .52-.87).
Change of preschoolers' sleep duration | Through study completion, 24 weeks
  Preschoolers' sleep duration will be assessed at baseline, at the end of 12-week post-intervention, and at the end of 12-week follow-up, using Garmin Vivofit Jr 3 Fitness Tracker for kids. According to the manufacturer, Vivofit Jr 3 can track sleep, as well as work as an alarm clock, timer, and watch. Vivofit can be placed in sleep mode to track sleep time, amount of restful sleep, and movement during sleep. The Vivofit data can be uploaded to a personal computer via a wireless USB ANT StickTM and viewed on the software created by the manufacturer.
Change of preschoolers' sleep problems | Through study completion, 24 weeks
  Children's sleep problems will be examined at baseline, at the end of 12-week post-intervention, and at the end of 12-week follow-up, using the Chinese version of the Children's Sleep Habits Questionnaire (CSHQ), which has been a frequently used parent survey to screen children aged from 4 to 10. It contains 33 items to form a different set of eight domains: bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night waking, parasomnia, sleep-disordered breathing, and daytime sleepiness. Each scored question is rated on a 3-point scale as "usually if something occurs 5 or more times in a week" (scored 3), "sometimes if something occurs 2-4 times in a week" (scored 2), "rarely if something occurs never or 1 time during a week" (scored 1). Higher scores represent greater sleep problems. The CSHQ has shown good reliability (Cronbach's Alpha is 0.73) and validity.
Change of parents' physical activity | Through study completion, 24 weeks
  Parent's PA will be assessed baseline, at the end of 12-week post-intervention, and at the end of 12-week follow-up, using the Chinese Version of the International Physical Activity-Long Form (IPAQ-L). The IPAQ-L has been shown to be a reliable and validated measure for assessing PA levels in Chinese cities.
Change of parenting style | Through study completion, 24 weeks
  Parenting style will be assessed baseline, at the end of 12-week post-intervention, and at the end of 12-week follow-up, using the Chinese version of parenting Style & Dimension Questionnaire, which is a self-report instrument designed to measure authoritarian (e.g., I yell when I disapprove of my child's behavior), authoritative (e.g., I am responsive to my child's feelings and needs), and permissive parenting style (e.g., I find it difficult to discipline my child) of 4-12 years old children's parents. This scale comprises 32 items, with each item of scale evaluated by the five points Likert described as "never", "once in a while", "about half of the time", "very often" and "always". The overall Cronbach Alpha is 0.87
Change of parenting feeding style | Through study completion, 24 weeks
  Parenting feeding style will be assessed baseline, at the end of 12-week post-intervention, and at the end of 12-week follow-up, using the Chinese Version of the Parent Feeding Style Questionnaire, which consists of 4 parts: instrumental feeding (4 items), emotional feeding (5 items), prompting or encouragement to eat (8 items), and control over eating (10 items). Respondents will be asked to choose from a 5-point Likert scale (ranging from "never" to "always"). For example, "I allow my child to choose which food to have for meals, I encourage my child to look forward to the meal." The average score on each scale will be calculated and a higher score indicated a greater tendency for parents to feed their children in that style. The overall Cronbach's Alpha is 0.75.

OTHER OUTCOMES:
Demographic information | Baseline
  Parents' information includes socioeconomic status (range of income, educational level, and occupational status), age, gender, marital status, and children's height, weight, birth order. (We will use SECA Medical Body Composition Analysis to measure Wight and Height. Weight is measured at 0.1 kg with the preschoolers barefoot and wearing light clothing and height is measured at 0.1 cm).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peng Z, Wen LM, Lau PWC. Effectiveness of a Parent-Based eHealth Intervention on Physical Activity, Dietary Behaviors, and Sleep in Preschoolers: Randomized Controlled Trial. J Med Internet Res. 2025 Sep 2;27:e70886. doi: 10.2196/70886. PMID 40896827
- [Derived] Peng Z, Lau PW, Wen LM. Moderating effects of demographic characteristics on the relationship between parenting practices and energy balance related behaviors of Chinese preschoolers. Front Public Health. 2024 Dec 24;12:1476733. doi: 10.3389/fpubh.2024.1476733. eCollection 2024. PMID 39776485
- [Derived] Zhou P, Song H, Lau PWC, Shi L, Wang J. Effectiveness of a Parent-Based eHealth Intervention for Physical Activity, Dietary Behavior, and Sleep Among Preschoolers: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Sep 12;13:e58344. doi: 10.2196/58344. PMID 39264108